CLINICAL TRIAL: NCT00288678
Title: A Prospective Study on Diabetes Management Through an Integrated Delivery System
Acronym: DMIDS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Responsible Party: Center for Healthy Policy Research and Development, National Health Research Institutes, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: HP-PP08
Record Dates: First submitted 2006-02-07; First posted 2006-02-08 (Estimated); Last update posted 2010-01-27 (Estimated); Status verified 2008-02

CONDITIONS: Diabetes Mellitus
Keywords: Diabetic shared care; Health manager; Prospective Study; Health Care Quality, Access, and Evaluation
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Health Education

SUMMARY:
1. To demonstrate a feasible hospital-based diabetic shared care model in Taiwan.
2. To compare effectiveness of diabetes control between patients receiving case management provided by a health manager and patients receiving usual care.
3. To determine the optimal level of glucose, blood pressure and lipids in control of diabetes in Taiwan.

DETAILED DESCRIPTION:
Five general hospitals, including both public and private, are chosen as regional coordinating centers in this project. Collaborating with community physicians, project coordinating-centers randomize diabetic patients, who have signed informed consent, into either intervention or control group. While two annual comprehensive lab tests are offered to the control group, an additional package of consultations and coordinating services provided by health managers is appended to the intervention group. Qualified health managers are cultivated in five selected medical institutes to support primary care physicians in managing diabetic patients. Responsibilities of health managers include tracking and updating enrolled patients' information, providing adequate and scheduled consultations, arranging specialty referrals for patients in needs, and transferring stable patients back to their original physicians. The feasibility phase of the project implementation will last for three years and it will be followed by a phase of full-scale implementation for another two years. Glycemic control as well as health status of participants will be the indicators to evaluate outcome of the project. At the same time, the periodic measurements on glucose, blood pressures, lipids and the incidence of complications will also be analyzed to set up an optimal target for diabetic control in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

1. Symptoms of diabetes plus casual plasma glucose concentration 200 mg/dl (11.1 mmol/l). Casual is defined as any time of day without regard to time since last meal. The classic symptoms of diabetes include polyuria, polydipsia, and unexplained weight loss.
2. Fasting plasma glucose 126 mg/dl (7.0 mmol/l). Fasting is defined as no caloric intake for at least 8 hours.

3.2-hour plasma glucose 200 mg/dl (11.1 mmol/l) during an oral glucose tolerance test (OGTT). The test should be performed using a glucose load containing the equivalent of 75-g anhydrous glucose dissolved in water.

Exclusion Criteria:

1. Type 1 diabetes (Insulin dependent diabetes, IDDM)
2. Women who are pregnant at the entry time.
3. Those who have history of myocardial infraction (MI), cerebrovascular accident (CVA), foot amputation and uremia under dialysis.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1222 (Actual)
Dates: Start 2003-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Through the health manager's coordination and consultation, diabetic patients will have better glycemic control for fasting plasma glucose, HbA1c, and blood cholesterol level.

SECONDARY OUTCOMES:
Patients in the intervention group will have better health status such as lower hospitalization rate, shorter length of stay in hospitals, and fewer diabetic complications.

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Cheng Hsu, M.D, Dr. P.H, Principal Investigator — National Health Research Instiutes; Hsing-Yi Chang, Ph. Dr. P.H, Principal Investigator — National Health Research Instiutes
Locations (5):
- Taiwan (5):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Tri-Services General Hospital, Taipei
  - Min-Shen General Hospital, Taoyuan District

REFERENCES:
- [Background] Harris MI, Flegal KM, Cowie CC, Eberhardt MS, Goldstein DE, Little RR, Wiedmeyer HM, Byrd-Holt DD. Prevalence of diabetes, impaired fasting glucose, and impaired glucose tolerance in U.S. adults. The Third National Health and Nutrition Examination Survey, 1988-1994. Diabetes Care. 1998 Apr;21(4):518-24. doi: 10.2337/diacare.21.4.518. PMID 9571335
- [Background] Lin T, Chou P, Lai MS, Tsai ST, Tai TY. Direct costs-of-illness of patients with diabetes mellitus in Taiwan. Diabetes Res Clin Pract. 2001 Nov;54 Suppl 1:S43-6. doi: 10.1016/s0168-8227(01)00308-4. PMID 11580968
- [Background] Chuang LM, Tsai ST, Huang BY, Tai TY; DIABCARE (Taiwan) Study Group. The current state of diabetes management in Taiwan. Diabetes Res Clin Pract. 2001 Nov;54 Suppl 1:S55-65. doi: 10.1016/s0168-8227(01)00310-2. PMID 11580970
- [Background] Chiou ST, Lin HD, Yu NC, Hseuh HK, Lin LH, Lin LT, Chen TJ, Lai MS. An initial assessment of the feasibility and effectiveness of implementing diabetes shared care system in Taiwan--some experiences from I-Lan County. Diabetes Res Clin Pract. 2001 Nov;54 Suppl 1:S67-73. doi: 10.1016/s0168-8227(01)00311-4. PMID 11580971
- [Background] Marshall CL, Bluestein M, Briere E, Chapin C, Darling B, Davis K, Davis T, Gersten J, Harris C, Hodgin A, Larsen W, Mabb D, Rigberg H, Watson D, Krishnaswami V. Improving outpatient diabetes management through a collaboration of six competing, capitated Medicare managed care plans. Am J Med Qual. 2000 Mar-Apr;15(2):65-71. doi: 10.1177/106286060001500205. PMID 10763220
- [Background] Mensing C, Boucher J, Cypress M, Weinger K, Mulcahy K, Barta P, Hosey G, Kopher W, Lasichak A, Lamb B, Mangan M, Norman J, Tanja J, Yauk L, Wisdom K, Adams C. National standards for diabetes self-management education. Task Force to Review and Revise the National Standards for Diabetes Self-Management Education Programs. Diabetes Care. 2000 May;23(5):682-9. doi: 10.2337/diacare.23.5.682. No abstract available. PMID 10834430
- [Background] Rubin RJ, Dietrich KA, Hawk AD. Clinical and economic impact of implementing a comprehensive diabetes management program in managed care. J Clin Endocrinol Metab. 1998 Aug;83(8):2635-42. doi: 10.1210/jcem.83.8.5075. PMID 9709924
- [Background] Chicoye L, Roethel CR, Hatch MH, Wesolowski W. Diabetes care management: a managed care approach. WMJ. 1998 Mar;97(3):32-4. PMID 9540446
- [Background] Expert Committee on the Diagnosis and Classification of Diabetes Mellitus. Report of the Expert Committee on the Diagnosis and Classification of Diabetes Mellitus. Diabetes Care. 2000 Jan;23 Suppl 1:S4-19. No abstract available. PMID 12017675
- [Background] American Diabetes Association. Standards of medical care for patients with diabetes mellitus. Diabetes Care. 2002 Jan;25(1):213-29. doi: 10.2337/diacare.25.1.213. No abstract available. PMID 11772918
- [Background] American Diabetes Association. Screening for type 2 diabetes. Diabetes Care. 2000 Jan;23 Suppl 1:S20-3. No abstract available. PMID 12017671
- [Derived] Huang MC, Chang WT, Chang HY, Chung HF, Chen FP, Huang YF, Hsu CC, Hwang SJ. FADS Gene Polymorphisms, Fatty Acid Desaturase Activities, and HDL-C in Type 2 Diabetes. Int J Environ Res Public Health. 2017 May 28;14(6):572. doi: 10.3390/ijerph14060572. PMID 28555039
- [Derived] Chung HF, Long KZ, Hsu CC, Al Mamun A, Jhang HR, Shin SJ, Hwang SJ, Huang MC. Association of n-3 polyunsaturated fatty acids and inflammatory indicators with renal function decline in type 2 diabetes. Clin Nutr. 2015 Apr;34(2):229-34. doi: 10.1016/j.clnu.2014.02.009. Epub 2014 Mar 19. PMID 24721145